CLINICAL TRIAL: NCT05564247
Title: Effectiveness of the Wheelchair Skills Training Program for Improving Wheelchair Skills and Related Rehabilitation Outcomes Among Children and Youth
Brief Title: Wheelchair Skills Training for Children and Youth
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WSP-Ped2021
Record Dates: First submitted 2022-06-14; First posted 2022-10-03 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Wheelchairs
Keywords: manual wheelchair; manual wheelchair skills training; pediatrics; self efficacy; skills capacity; skills performance; satisfaction with participation; actigraphy

STUDY DESIGN:
Intervention Model Description: A three-site, single-blind randomized controlled trial (RCT)
Who Masked: Participant, Care Provider
Masking Description: Testers will remain blinded to group assignment throughout the study. A Research Coordinator (Quebec site) will coordinate T2 and T3 assessments for both groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (WSTP) (Experimental): Participants will complete 12, 45-minute weekly sessions of WSTP delivered by clinicians with >5 years of experience working with children who use MWC. Trainers will customize each session based on the age group (child or adolescent) and training goals of each child as determined in session one. Subsequent sessions will begin with a 5-minute review of progress and socializing, followed by a 10-minute warm-up (random practice of the previously learned skills); 20 minutes of attempting new skills (training on each skill will be carried to next session until the skills are learned or until the trainer and participant mutually agree that training should be abandoned; the trainer will periodically ask the participant to practice newly learned skills to incorporate variability of practice); 10 minute cool-down, during which the participant will practice skills in a self-controlled environment. Age-appropriate considerations are incorporated into training materials
  Interventions: Behavioral: Wheelchair Skills Training Program (WSTP)
- Control Group (Attention) (No Intervention): Participants will be attention-matched to mimic time and contacts ‬of‭ ‬the‭ experimental‭ ‬group. The control group will receive 12, 45-minute weekly sessions of 'Games and Activities' facilitated by healthcare professionals (e.g., occupational therapy/rehabilitation students) who will not be involved in the intervention or any other aspect of the study. The control group facilitator will mimic the same type of attention as the training at each site (i.e., sessions will be held at healthcare facilities and in the community (e.g., libraries, shopping centres, museums, parks). Facilitators will be equipped with current popular games and activities (according to social media and websites of popular children's stores) kits that include various board and card games, hand-eye coordination games, active games, cognitive activities, and arts and crafts suitable for children and adolescents to ensure interest and acceptability for all participants.

INTERVENTIONS:
Behavioral: Wheelchair Skills Training Program (WSTP) — Participants will complete customized MWC skills training based on the evidence-based wheelchair skills program. Lessons plans will be created by the clinicians, children and parents participants based on goals, age, skills and interests, and used to customize the training.
  Arms: Experimental Group (WSTP)

SUMMARY:
Manual wheelchair (MWC) skills training is a critical component of wheelchair service provision. However, children and youth receive little to no training. MWC training effectively improves MWC skills, self-efficacy and satisfaction with participation (ie., facilitators of independent mobility and social participation) in adults. Independent mobility is especially critical for children, as it is associated with higher likelihood of employment and independent living in adulthood.

Despite evidence of an effective Wheelchair Skills Training Program (WSTP) for adults, very little research has been conducted in the area of wheelchair mobility for children and youth. Two small single-group studies suggest that MWC skills training improves wheelchair skills and satisfaction with participation among individuals ages 4-17 years when training was conducted by professionals (eg. clinicians) and non-professionals (eg. peer-trainers). However, there are no controlled trials documenting the effect of MWC skills training among children and no evidence of best training approaches.

The purpose of this study is to evaluate the efficacy of the WSTP for improving MWC skills, MWC confidence and participation outcomes among children and youth. A randomized controlled trial will establish efficacy of clinician led approaches to training, which may be implemented on a broader community-based scale in the future.

The results of this study will provide critical evidence for best practices for improving MWC mobility during childhood. Deliverables from this study will include MWC skills training tools for clinicians, that will be made freely available through an existing website. The results will support multi-site implementation trials and exploration of community-based approaches to wheelchair skills training for children and use.

DETAILED DESCRIPTION:
Goal. Evaluate the efficacy of the Wheelchair Skills Training Program (WSTP) (ie. the current gold-standard among adults) for improving MWC skills (primary outcome), MWC activity, MWC use self-efficacy, satisfaction with participation, among children and youth ages 4 to 21 years. The influence of the WSTP on parents perception of their child's MWC skills and parent's satisfaction with participation will also be evaluated.

Background: Manual wheelchair (MWC) skills training is a critical component of service provision. Sixteen randomized controlled trials (RCTs) and two meta-analyses demonstrate that a Wheelchair Skills Training Program (WSTP) effectively improves MWC skills among adults. Evidence also suggests that the WSTP can improve self-efficacy for using a MWC and satisfaction with participation (ie. facilitators of independent mobility and social participation). Among children and youth (5-17 years), two quasi-experimental trials have shown improved wheelchair skills and satisfaction with participation when the WSTP was conducted by both professionals (eg. occupational therapists, physiotherapists) and non-professionals (eg. peer-trainers). To date there are no experimental trials evaluating the efficacy of MWC skills training among children and youth, and there is limited evidence on the best approach to training.

Research aims: The purpose is to evaluate the efficacy of the WSTP, for improving wheelchair skills (primary outcome), parent-perceived wheelchair skills, satisfaction with participation in meaningful activities, wheelchair use self-efficacy, and health-related quality of life among children and youth, compared to usual wheelchair training practice, and to measure the retention of benefits 6 months later.

Methods: A 3-site (Quebec City, Montreal, Halifax) RCT will be conducted in both official languages. Forty-eight children and youth ages 4-21 years will be randomized (stratified by site and by age groups {ie. 4-7, 8-11, 12-16, and 17-21}) to the intervention group or control group. The intervention group will receive 10 sessions of the WSTP (modified for children and youth) facilitated by healthcare professionals (e.g., occupational therapists, physiatrists). The control group will receive an attention control and usual wheelchair provision and services at each site. Between-group analysis will be conducted with primary (wheelchair skills) and secondary outcomes (parent-perceived wheelchair skills, satisfaction with participation, self-efficacy and health-related quality of life and a 6-month follow-up will be conducted. Qualitative interviews will explore experiential aspects of participation.

Core expertise. World leaders in wheelchair skills training (ie, developers of the WSTP) form this pan-Canadian interdisciplinary team. The study team has expertise in administering the WSTP and all outcomes in English and French, implementation of multi-site RCTs, and recruitment of wheelchair users. Clinical and community collaborators are interested in adopting the WSTP for use in child and youth populations and have committed their support to this project.

Expected outcomes: Demonstrating the efficacy of the WSTP for children and youth will provide an evidence-based program that is ready for uptake by healthcare professionals and possibly scalable for community-based professionals and non-professionals across Canada and the world. Working with clinical and community partners will position us to negotiate knowledge dissemination and sustainability of an efficacious program. The WSTP may improve independent mobility, confidence and participation outcomes in children and youth of various ages, while reducing risk of injury and burden on parents and families. Independent mobility during childhood is associated with higher likelihood of employment and independent living in adulthood.

ELIGIBILITY:
Inclusion Criteria:

* have their own Manual Wheelchair (MWC)
* able to self-propel MWC for a minimum distance of 10 metres, without assistance
* able to follow a two-step command (evaluated by person conducting eligibility screening)

Exclusion Criteria:

* anticipate health conditions/procedures that contraindicate training in the next 6 months (e.g. surgery)
* have a degenerative condition that is expected to progress quickly
* will be/ are attending MWC skills training

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-07-24 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Wheelchair Skills Test Version 5.3.1 for MWC users | Baseline (T1); immediately post intervention up to 12 weeks after baseline (T2); 6-months follow-up (T3)
  Change in MWC skills capacity (i.e., what a person can do in a standardized environment), and frequency of performance will be assessed using the Wheelchair Skills Test (WST). Each item is scored on a scale from 0 to 3, with 0= not capable to perform the skill (or not safely), 1 = can perform the skill partially; 2= can perform the skill (but has room for improvement); 3= can perform the skill at an expert level. A percent score is calculated, with higher percentage = higher skills.

SECONDARY OUTCOMES:
Manual Wheelchair Activity (Actigraph) | Baseline (T1); immediately post intervention up to 12 weeks after baseline (T2); 6-months follow-up (T3)
  Change in objective MWC activity will be collected to triangulate measurement of improvement in MWC skills and engagement in community activities using a triaxial accelerometer (Actigraph GT3X, Pensacola FL).
Parents Perception of Child's MWC Capacity and Performance Version 5.2.1 | Baseline (T1); immediately post intervention up to 12 weeks after baseline (T2); 6-months follow-up (T3)
  Change in parents' ratings of their child's performance each of the 33 skills on the Wheelchair Skills Test-Questionnaire. Each item is scored on a scale from 0 to 3, with 0= not capable to perform the skill (or not safely), 1 = can perform the skill partially; 2= can perform the skill (but has room for improvement); 3= can perform the skill at an expert level. A percent score is calculated, with higher percentage = higher skills.
MWC Use Confidence Scale (Wheel use confidence scale) | Baseline (T1); immediately post intervention up to 12 weeks after baseline (T2); 6-months follow-up (T3)
  Change in perceived self-efficacy for wheelchair use is rated on a 33-item scale, where children rate their level of confidence on a scale from 0 to 10. Each item is scored on a scale from 0 to 10, with 0= not confident at all, 10 = very confident. A percent score is calculated. Higher percentage = higher confidence.
The Wheelchair Outcome Measure for Young People (WhOM-YP) | Baseline (T1); immediately post intervention up to 12 weeks after baseline (T2); 6-months follow-up (T3)
  Change in ratings of satisfaction with social participation and activity performances in a wheelchair is evaluated using a semi-structured questionnaire, in which participants identify personal goals that require the use of a wheelchair (e.g., preparing meals, playing with friends at school). Parents and children can each develop up to 5 indoor goals and 5 outdoor goals. Each goal is rated for level of importance (scale from 0 to 10) and level of satisfaction (scale from 0 to 10). Importance and frequency scores are multiples to give a score out of 100, and an average score is calculated with the denominator dependent on the number of goals. A percentage score is calculated with higher scores indicative of higher satisfaction with goal attainment.

CONTACTS AND LOCATIONS:
Overall Officials: Krista Best, PhD, Principal Investigator — Universite Laval
Locations (3):
- Canada (3):
  - IWK Health Centre, Halifax, Nova Scotia
  - CHU Ste-Justine, Montreal, Quebec
  - Universite Laval, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Best KL, Rushton PW, Sheriko J, Arbour-Nicitopoulos KP, Dib T, Kirby RL, Lamontagne ME, Moore SA, Ouellet B, Routhier F. Effectiveness of wheelchair skills training for improving manual wheelchair mobility in children and adolescents: protocol for a multicenter randomized waitlist-controlled trial. BMC Pediatr. 2023 Sep 26;23(1):485. doi: 10.1186/s12887-023-04303-8. PMID 37752480